CLINICAL TRIAL: NCT05377528
Title: A Phase 1 Study Investigating AGEN1571 as a Single Agent and in Combination With a PD-1 Inhibitor and/or Botensilimab (AGEN1181) in Patients With Advanced Solid Tumors
Brief Title: Study of AGEN1571 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C-1500-01
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Cancer; Open-label; Dose Escalation; Dose Expansion; Monotherapy; Combination Therapy; Anti-CTLA-4; Anti-PD-1; ILT2
MeSH Terms: interventions — balstilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation: AGEN1571 (Experimental): Participants will receive AGEN1571 monotherapy.
  Interventions: Drug: AGEN1571
- Dose Escalation: AGEN1571 + Balstilimab (Experimental): Participants will receive AGEN1571 with balstilimab.
  Interventions: Drug: AGEN1571; Drug: Balstilimab
- Dose Escalation: AGEN1571 + Botensilimab (Experimental): Participants will receive AGEN1571 with botensilimab.
  Interventions: Drug: AGEN1571; Drug: Botensilimab
- Dose Escalation: AGEN1571 + Balstilimab + Botensilimab (Experimental): Participants will receive AGEN1571 with balstilimab and botensilimab.
  Interventions: Drug: AGEN1571; Drug: Balstilimab; Drug: Botensilimab
- Dose Expansion (Experimental): AGEN1571 administered at the RP2D for monotherapy or any combination therapy.
  Interventions: Drug: AGEN1571; Drug: Balstilimab; Drug: Botensilimab

INTERVENTIONS:
Drug: AGEN1571 — A fully human monoclonal immunoglobulin-like transcript antagonist antibody administered intravenously.
Drug: Balstilimab — A fully human monoclonal programmed cell death protein 1 antagonist antibody administered intravenously.
  Other Names: AGEN2034
  Arms: Dose Escalation: AGEN1571 + Balstilimab; Dose Escalation: AGEN1571 + Balstilimab + Botensilimab; Dose Expansion
Drug: Botensilimab — A fully human fragment crystallizable-enhanced monoclonal cytotoxic T lymphocyte antigen 4 antibody administered intravenously.
  Other Names: AGEN1181
  Arms: Dose Escalation: AGEN1571 + Balstilimab + Botensilimab; Dose Escalation: AGEN1571 + Botensilimab; Dose Expansion

SUMMARY:
This is an open-label, Phase 1, 2-part trial to determine recommended phase 2 doses (RP2Ds) and evaluate the safety, tolerability, pharmacokinetic, and pharmacodynamic profiles of AGEN1571 both as a monotherapy and in combination with balstilimab (PD-1 inhibitor) and/or botensilimab (2-agent combination or 3-agent combination) in participants diagnosed with advanced solid tumors.

Part 1 will be the dose escalation phase to determine the RP2D of AGEN1571 monotherapy or AGEN1571 in combination with balstilimab and/or botensilimab. Part 2 will be the dose expansion phase for specific disease indications. Participants will receive study treatment for up to 2 years, or until any disease progression, unacceptable toxicity, or participant wishes to withdraw consent for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate by giving signed, dated, and written informed consent prior to any study-specific procedures (participation in genetic testing is optional).
2. Histologically confirmed diagnosis of a solid tumor that is currently metastatic or locally advanced for which no standard therapy is available or standard therapy has failed.
3. Measurable disease on baseline imaging based on RECIST 1.1.
4. Life expectancy of at least 3 months.
5. Eastern Cooperative Oncology Group performance status of 0 or 1.
6. Adequate organ and bone marrow reserve function, as indicated by the following laboratory values:

   1. Adequate hematological function, defined as absolute neutrophil count ≥ 1.5 × 10^9/liter (L), platelet count ≥ 100 × 10^9/L, and hemoglobin ≥ 8 grams (g)/deciliter (dL) without recent transfusion (defined as a transfusion that has occurred within 2 weeks of the hemoglobin measurement).
   2. Adequate liver function, defined as serum albumin ≥ 3.0 g/dL, total bilirubin level ≤ 1.5 × institutional upper limit of normal (IULN), aspartate aminotransferase ≤ 2.5 × IULN, and alanine aminotransferase ≤ 2.5 × IULN, and alkaline phosphatase ≤ 2.5 × IULN or ≤ 5 × IULN for participants with liver metastases.
   3. Adequate renal function defined as calculated creatinine clearance ≥ 40 milliliters/minute as assessed by Cockcroft-Gault method.
   4. Adequate coagulation, defined as international normalized ratio or prothrombin time ≤ 1.5 × IULN and activated partial thromboplastin time ≤ 1.5 × IULN (unless participant is receiving anticoagulant therapy).
7. Participants with a history of prior malignancy are eligible if treatment was completed ≥ 2 years prior to the first dose of study treatment and the participant has no evidence of disease. Participants who have been maintained on stable doses of antineoplastic hormonal therapy within that 2-year time frame may also be eligible with approval of the Medical Monitor. Participants with a history of prior early-stage basal/squamous cell skin cancer, or noninvasive or in situ cancers, who have undergone definitive treatment at any time are also eligible.
8. Participants must provide a sufficient and adequate formalin-fixed paraffin embedded tumor tissue sample (biopsy) collected after the last dose of prior anti-cancer therapy and before the first dose of study treatment from a site not previously irradiated and agree to a mandatory on-treatment biopsy, if clinically feasible. If a potential study participant cannot provide a tumor tissue sample as specified above, enrollment may be possible following discussion and approval from the Medical Monitor.
9. Female participants of childbearing potential must have a negative urine or serum pregnancy test at screening (within 72 hours of first dose of study medication) with repeat urine or serum pregnancy test on Day 1 of each cycle and at the End of Treatment visit. If a urine pregnancy test is positive, results must be confirmed with a serum pregnancy test. Non-childbearing potential is defined as follows:

   1. ≥ 50 years of age and has not had menses for greater than 1 year.
   2. Amenorrheic for ≥ 2 years without a hysterectomy and bilateral oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation.
   3. Status is post hysterectomy, bilateral oophorectomy, or tubal ligation.

   Female participants who are diagnosed with a tumor that is known to secrete human chorionic gonadotropin must be certified not pregnant based on clinical evidence and investigator judgment.

   Female participants of child-bearing potential must agree to use highly effective contraceptive measures starting with the screening visit through 90 days after the last dose of study treatment.

   Note: Abstinence is acceptable if this is the established and preferred contraception for the participant.
10. Male participants with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study starting with the screening visit through 90 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

    Note: Abstinence is acceptable if this is the established and preferred contraception for the participant.
11. Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of first dose of current study drug.
2. Received prior systemic cytotoxic chemotherapy, biological therapy, radiotherapy, or major surgery outside of the acceptable washout periods prior to first dose of study drug. The following washout windows are acceptable from prior treatments, that is participants with time periods less than the following should be excluded:

   1. Cytotoxic agent or monoclonal antibody ≥ 3 weeks is acceptable (that is, < 3 weeks should be excluded).
   2. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease.
   3. Small molecule targeted investigational therapies and tyrosine kinase inhibitors ≥ 14 days or 5 half-lives is acceptable (that is, < 14 days or < 5 half-lives should be excluded).
   4. Having a previous severe acute respiratory syndrome coronavirus 2 vaccine > 7 days before administration is acceptable. For vaccines requiring more than 1 dose, the full series should be completed prior to Cycle 1 Day 1 (C1D1), when feasible, and when the delay in initiation of study treatment would not put the study participants at risk.
   5. Prior radiation therapy to the CNS within 2 weeks before first treatment.
3. Persistent toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 Grade >1 severity that is related to prior therapy.

   a. Sensory neuropathy or alopecia of Grade ≤ 2 is acceptable. Stable, compensated endocrinopathies (hypothyroidism, adrenal insufficiency, hypophysitis) that are the sequelae of immune-mediated adverse events > Grade 1 are acceptable.
4. Known severe (Grade ≥ 3) hypersensitivity reactions to fully human monoclonal antibodies, or to any study drug excipients, or severe reaction to immuno-oncology agents, such as colitis or pneumonitis requiring treatment with steroids; or has a history of or active interstitial lung disease, any history of anaphylaxis, or uncontrolled asthma.
5. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 milligrams [mg] daily prednisone equivalent) within 14 days or any other immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses (≤ 10 mg daily prednisone equivalent), are permitted in the absence of active autoimmune disease.
6. Active CNS metastases. Note: Participants are eligible if CNS metastases have been treated and participants are radiologically and clinically stable. Participants must have been either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone or equivalent for at least 2 weeks prior to the first dose of study treatment.
7. Active or history of autoimmune disease that requires systemic treatment within 2 years of the start of study drug (that is, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Note: Participants with autoimmune conditions requiring hormone replacement therapy or topical treatments are eligible.
8. Participants has had an allogeneic tissue/solid organ transplant, except for corneal transplants.
9. An active infection requiring treatment within 2 weeks of C1D1, or active interstitial lung disease.
10. Human immunodeficiency virus (HIV) positive:

    1. Participants with cluster of differentiation 4 > 200 cells/cubic millimeter are eligible.
    2. Participants with undetectable HIV viral load are eligible.
11. Active hepatitis B (HBV) or active hepatitis C (HCV).

    1. Participants with HBV infection are eligible if HBV surface antigen and HBV DNA are negative.
    2. Participants with HCV infection are eligible if HCV RNA is negative.
12. Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication.
13. History or current evidence of any condition (including psychiatric or substance abuse disorder that would interfere with the requirements of the trial), therapy, any active infection requiring treatment within 2 weeks of C1D1, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
14. Legally incapacitated or has limited legal capacity.
15. Pregnant or breastfeeding.
16. Corrected QT interval (QTc) > 480 milliseconds at screening except if the prolonged QTc is due to right bundle branch block.
17. Uncontrolled hypertension or controlled hypertension (> 140/90 millimeters of mercury) on more than 3 antihypertensive agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Number Of Participants With Dose-limiting Toxicities | Day 1 through Day 42
Number Of Participants With Treatment-emergent Adverse Events | Day 1 up to 12 months after the last dose

SECONDARY OUTCOMES:
Serum AGEN1571 Concentration | Day 1 up to 90 days after the last dose
Serum Balstilimab Concentration | Day 1 up to 90 days after the last dose
Serum Botensilimab Concentration | Day 1 up to 90 days after the last dose
Number Of Participants With Anti-drug Antibodies | Day 1 up to 90 days after the last dose
Overall Response Rate (ORR) | Day 1 up to 90 days after the last dose
  ORR will be determined using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Complete Response (CR) Rate | Day 1 up to 90 days after the last dose
  CR will be determined using RECIST 1.1.
Partial Response (PR) Rate | Day 1 up to 90 days after the last dose
  PR will be determined using RECIST 1.1.
Duration Of Response (DOR) | Day 1 up to 90 days after the last dose
  DOR will be determined using RECIST 1.1.
Disease Control Rate (DCR) | Day 1 up to 90 days after the last dose
  DCR will be determined using RECIST 1.1.
Progression-free Survival (PFS) | Day 1 up to 90 days after the last dose
  PFS will be determined using RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Lifespan Cancer Institute, Providence, Rhode Island